CLINICAL TRIAL: NCT04052178
Title: Sensory Neuromodulation Protocol for the Treatment of Post-stroke Oropharyngeal Dysphagia. Short-term Neurophysiological Effects.
Brief Title: Sensory Neuromodulation Protocol for the Treatment of Post-stroke Oropharyngeal Dysphagia.
Acronym: FIS2014
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Mataró (Other)
Responsible Party: Principal Investigator, Pere Clave, Academic Director of Research and Development of the Hospital de Mataró, Hospital de Mataró
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FIS2014
Record Dates: First submitted 2019-08-02; First posted 2019-08-09 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Swallowing Disorder; Dysphagia; Stroke; Neurophysiologic Abnormality
Keywords: Oropharyngeal dysphagia; Stroke; Sensory stimulation
MeSH Terms: conditions — Deglutition Disorders; Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Repetitive transcranial magnetic stimulation (rtMS) (Active Comparator): Acute repetitive transcranial magnetic stimulation on the pharyngeal sensory cortex. Applied intensity 90% of the resting motor threshold, 1250 pulses at 5 Hz.
  Each treatment arm was placebo/sham compared with a time separation of one week. The assignment to either active or sham was randomized.
  Interventions: Device: rTMS active and sham
- Intrapharyngeal electrical stimulation (PES) (Active Comparator): Intrapharyngeal electrical stimulation applied to an intensity of 75% of the tolerance threshold with 0.2 ms pulses at 5 Hz during 10 min.
  Each treatment arm was placebo/sham compared with a time separation of one week. The assignment to either active or sham was randomized.
  Interventions: Device: PES active and sham
- Capsaicin (Active Comparator): 100 mL of oral capsaicin solution at a concentration of 10-5M.
  Each treatment arm was placebo/sham compared with a time separation of one week. The assignment to either active or sham was randomized
  Interventions: Dietary Supplement: Capsaicin active and placebo

INTERVENTIONS:
Device: rTMS active and sham — Repetitive transcranial magnetic stimulation of the pharyngeal sensory cortex.
  Other Names: Repetitive transcranial magnetic stimulation
  Arms: Repetitive transcranial magnetic stimulation (rtMS)
Device: PES active and sham — Intrapharyngeal electrical stimulation with a catheter delivering electrical pulses.
  Other Names: Intrapharyngeal electrical stimulation
  Arms: Intrapharyngeal electrical stimulation (PES)
Dietary Supplement: Capsaicin active and placebo — Capsaicin solution (TRPV1 agonist) at a concentration of 10-5M or placebo solution.
  Other Names: TRPV1 agonist (capsaicin at 10-5M) or placebo
  Arms: Capsaicin

SUMMARY:
Study design: Multicenter, experimental, randomized, crossed, double blind study (patient and results analysis).

Aim: To evaluate the effect of different neurostimulation techniques on the neurophysiological and biomechanical swallowing mechanisms of patients with dysphagia associated with chronic stroke and select those techniques with the best results to be evaluated in the second phase of the study (medium-term effects).

Outcome measures:

* Videofluoroscopy: prevalence of impaired efficacy and safety of swallow (penetrations and aspirations), penetration aspiration scale (PAS: from 0 to 8), biomechanical parameters (time to laryngeal vestibule closure, upper esophageal sphincter opening).
* Pharyngeal sensory evoked potentials (pSEP): latency and amplitude of obtained evoked potentials. Higher latency (0 onwards) means worse outcome and higher amplitude (0 onwards) means better outcome.
* Pharyngeal motor evoked potentials (pMEP): latency, amplitude, duration and area of obtained evoked potentials. Higher latency (0 onwards) means worse outcome and higher amplitude (0 onwards) means better outcome.

Treatments and patients: 36 post-stroke patients with oropharyngeal dysphagia (PAS superior or equal to 2) randomized patients in 3 treatment arms (3 groups of 12 patients).

* Active and sham repetitive transcranial magnetic stimulation (rTMS): 90% of the resting motor threshold, 1250 pulses, 5 Hz.
* Active and sham Intrapharyngeal Electrical Stimulation (PES): 75% of tolerance threshold, pulses of 0.2 ms, 5 Hz, 10 min.
* Oral Capsaicin (active intervention, 10-5M, TRPV1 agonist) and placebo solution (sham): 100 mL, single administration.

Administration of study therapies:

The study will be performed in two visits separated for one week. In each visit patients will randomly receive active or sham treatment and a pre-post evaluation of biomechanics of deglutition (with VFS) and neurophysiological mechanisms (swallowing afferent and efferent pathways) will be performed in each visit.

Acute randomized administration -> 1 active session (pre/post evaluation with VFS/pSEP/pMEP) + 1 separate control session 1 week apart (pre/post evaluation with VFS/pSEP/pMEP).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Patients with a diagnosis of stroke of more than 3 months of evolution.
* Patients with clinical signs of dysphagia according to the volume viscosity swallowing test (V-VST).
* Patients capable of complying with the study protocol.
* Explained study and signed informed consent.

Exclusion Criteria:

* History of severe neurodegenerative, digestive diseases, epilepsy or previous seizures.
* Pacemaker or implanted defibrillator carriers.
* Implanted electrode carriers or other stimulation systems.
* Implant carriers or metal plates on the head or neck.
* Cochlear implant carriers.
* Medication pump carriers.
* History of hearing loss associated with noise.
* Cardiopulmonary instability.
* Oropharyngeal dysphagia of structural causes.
* History of head and neck surgery.
* Alcohol or drug dependence.
* Pregnancy or breastfeeding.
* Participate or have participated in another clinical interventionist trial in the 4 weeks prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Pharyngeal motor evoked potential (pMEP): latency and amplitude | The event wil be assessed with pMEP immediately after the application of the intervention (time frame maximum up to 2 hours).
  Study the magnitude of the effect by calculating the change of the evoked potential from baseline immediately after the application of the intervention produced by the different treatments. This will be examined and compared between active and sham intervention.
Pharyngeal sensory evoked potential (pSEP): latency and amplitude | The event wil be assessed with pSEPs immediately after the application of the intervention (time frame maximum up to 2 hours).
  Study the magnitude of the effect by calculating the change of the evoked potential from baseline immediately after the application of the intervention produced by the different treatments. This will be examined and compared between active and sham intervention.
Penetration-aspiration scale (PAS) score | The event wil be assessed with the PAS score immediately after the application of the intervention (time frame maximum up to 2 hours from first assessment).
  Study the magnitude of the effect by calculating the change on the prevalence of unsafe swallow (PAS≥2) in videofluoroscopy (VFS) from baseline immediately after the application of the intervention. This will be examined and compared between active and sham intervention.

SECONDARY OUTCOMES:
Opening and closing time of the laryngeal vestibule | The event wil be assessed with VFS immediately after the application of the intervention (time frame maximum up to 2 hours from first assessment).
  Time of the laryngeal vestibule opening and closure ranges from 0 to 1000 ms.
Prevalence of pharyngeal residue | The event will be assessed with VFS immediately after the application of the intervention (time frame maximum up to 2 hours from first assessment).
  The presence of pharyngeal residue in individual subjects will be assessed.
Resting motor threshold (RMT) of the pharyngeal cortex | The event wil be assessed with TMS immediately after the application of the intervention (time frame maximum up to 2 hours from first assessment).
  RMT is defined as the stimulation intensity in which the half of the stimuli are able to evoke a motor evoked potential of al least 10 uV of amplitude.
Pharyngeal sensory thresholds | The event wil be assessed with pharyngeal electrical stimulation immediately after the application of the intervention (time frame maximum up to 2 hours from first assessment).
  First perception and tolerance thresholds (from 0 to 100 mA) to electrical stimulation of the pharynx will be assessed by asking subjects the exact moment of first perception of the stimulus and the moment in which stimulation is not further tolerated, respectively.
Incidence of Treatment-Emergent Adverse Events | Although its occurrence is early after the TMS session, seizures and other side effects will be monitored up to 3 months after the intervention.
  Seizures are the most feared side effect associated with transcranial magnetic stimulation (TMS). Seizures are a rare side event during and/or subsequent to a TMS session (1.4%, Bae et al., 2007) commonly not occurring beyond a few days after the last session. No other major or significant side effects are expected associated with the interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Pere Clavé, PhD, Principal Investigator — Hospital de Mataró

IPD SHARING:
Plan to Share IPD: No